CLINICAL TRIAL: NCT06157515
Title: Inhaled Dose Analysis Using a Breath Actuated Nebulizer in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: National Tsing Hua University (Other); Chang Gung Memorial Hospital (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hui-Ling Lin, Professor, Department of Respiratory Therapy, Chang Gung University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: BANinHealthy
Record Dates: First submitted 2023-11-25; First posted 2023-12-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers; Aerosol Therapy; Inhaled Drug Dose; Pharmacogenomic Drug Interaction
Keywords: Vibrating Mesh Nebulizer; Breath-actuated Nebulization

STUDY DESIGN:
Intervention Model Description: This is a prospective crossover interventional study comparing two vibrating mesh nebulizer modalities - continuous versus breath-actuated - for delivering a bronchodilator, tested in healthy adult volunteers. Participants will receive an approved therapeutic dosage (2.5 mg salbutamol) via both devices in an alternating sequence. Outcome measurements focus on pharmacokinetic results, specifically urinary drug recovery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous vibrating mesh nebulization (cVMN) (Experimental): Participants will inhale 2.5 mg salbutamol (from a 0.5 unit dose vial of Saldolin Inhalation Solution, Taiwan FDA approval number 043572) via the commercially available vibrating mesh nebulizer (Microbase, model number MBPN002). The device continuously generates aerosol throughout the respiratory cycle. Participants are encouraged to breathe with normal tidal breathing for up to 5 minutes until no aerosol is visually seen. No repeat or additional dosing is utilized.
  Interventions: Device: Continuous vibrating mesh nebulizer
- Breath-actuated vibrating mesh nebulizer (bVMN) (Experimental): Participants will inhale 2.5 mg salbutamol (from a 0.5 unit dose vial of Saldolin Inhalation Solution, Taiwan FDA approval number 043572) via the commercially available vibrating mesh nebulizer (Microbase, model number MBPN002) with trigger module attachment. This device utilizes a microphone and algorithm to detect the inspiration to activate aerosol generation during period of inspiration only. Participants are encouraged to breathe with normal tidal breathing for up to 5 minutes until no aerosol is visually seen. No repeat or additional dosing is utilized.
  Interventions: Device: Breath-actuated vibrating mesh nebulizer

INTERVENTIONS:
Device: Breath-actuated vibrating mesh nebulizer — The intervention utilizes a breath-actuated vibrating mesh nebulizer system consisting of a controller module with microphone for respiratory phase detection and algorithm for inspiration triggering. This interfaces with the vibrating mesh nebulizer module which incorporates a micro-pump chip using piezoelectric effects to eject fluid through a mesh aperture plate holes. By detecting the onset of inspiration based on characteristic acoustic patterns using machine learning models, the controller module sends signals activating the piezoelectric vibration mechanism to generate aerosol only during the inspiratory phase through precision timing control, shutting off mist during expiration. The core module is attached to a standard commercial vibrating mesh nebulizer using the standard adult reusable mouthpiece interface.
  Other Names: Microbase, Model Number MBPN002 with trigger system
  Arms: Breath-actuated vibrating mesh nebulizer (bVMN)
Device: Continuous vibrating mesh nebulizer — When the continuous vibrating mesh nebulizer powered on, the micro-pump chip provides sustained vibrations onto the aperture plate, forcing fluid through micron-scale pores under pressure to continuously produce aerosol throughout inspiration and expiration phase.
  Other Names: Microbase, Model Number MBPN002
  Arms: continuous vibrating mesh nebulization (cVMN)

SUMMARY:
The goal of this crossover study is to compare urine drug concentrations using a continuous vibrating mesh nebulizer versus a breath-actuated vibrating mesh nebulizer in healthy volunteers. The main questions it aims to answer are:

* Whether breath-actuation nebulizer delivers higher inhaled drug dose, resulting in higher urine drug concentrations compared to continuous nebulization.
* Whether the different nebulizer modes deliver inhaled drug resulting in different effects on physiological parameters, including heart rate, respiratory rate, blood pressure, and blood oxygen saturation.

Participants will

* Inhale one dose (2.5mg) of salbutamol via continuous vs. breath-actuated nebulize mode.
* collect urine samples at multiple timepoints before and after nebulization to quantify drug elimination.

Researchers will compare the continuous and breath-actuated modes of vibrating mesh nebulizers to determine if breath-actuation improves drug delivery efficiency compared to continuous nebulization.

DETAILED DESCRIPTION:
Study Design and Objectives

This is a crossover study comparing two different nebulizer modes: continuous vibrating mesh nebulizer (cVMN, Microbase Inc.) vs. breath-actuated vibrating mesh nebulizer (bVMN, Microbase plus an actuated system) for bronchodilator delivery in 30 healthy volunteers. The primary objective is to compare urinary drug concentrations after inhalation between the two nebulizer modes to confirm an equivalent inhaled dose. Secondary objectives is to evaluate device safety based on vital sign changes and compare environmental drug particle concentrations between nebulizer modes.

Endpoints

The primary pharmacokinetic endpoint is urinary drug (salbutamol) concentration over 24 hours following nebulization with each mode. Secondary endpoints include pre- and post-nebulization vital signs (heart rate, blood pressure, respiratory rate, Saturation).

Study Procedures

Participants meeting the eligibility criteria will be assigned either to the continuous vibrating mesh nebulizer (cVMN) or the breath-actuated vibrating mesh nebulizer (bVMN). At visit 1, a baseline urine sample will be collected, followed by nebulization with a 0.5-unit dose (2.5 mg/1.25 mL salbutamol). Participants will inhale with normal tidal breathing for up to 5 minutes until the aerosol is visually seen. Vital signs will be continuously monitored every 5 minutes until 30 minutes after nebulization. Environmental particle concentration will be continuously measured by an aerosol spectrometer. Urine samples will be obtained 30 minutes before, 30 minutes after, and 24 hours post-nebulization. Visit 2 will follow identical procedures with the alternate nebulizer mode after a 1-week washout period.

Device Details

The cVMN is a commercially available continuous vibrating mesh nebulizer registered with the Taiwan Food and Drug Administration (device number 004561). The bVMN system incorporates a proprietary trigger module to enable breath-actuated delivery synchronized during inspiration. This module includes microphone detection during inspiration and expiration phases, along with software control of nebulization activation. Both devices utilize the same core nebulizer hardware and mesh component for aerosol generation.

Data Collection and Statistics

Urine samples will be extracted and analysis by HPLC to quantify salbutamol levels. Statistical analysis will include paired t-tests or nonparametric tests as appropriate to compare pharmacokinetic parameters, environmental concentrations, and vital signs changes between the two nebulize modes. Linear regression will also correlate urinary drug levels with nominal dose. The level of significance will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a written informed consent form.
* Healthy male and female participants aged >20 years.
* Forced expiratory volume in the first second (FEV1) greater than 80% of the predicted value.

Exclusion Criteria:

* Pregnant or lactating women.
* Regular use of bronchodilators or inhaled medications.
* History of bronchodilator allergy.
* Hyperthyroidism.
* Diabetes.
* History of heart disease.
* Arrhythmia.
* Angina.
* Hypertension.
* History of glaucoma, hypokalemia, or hyperglycemia.
* Severe anemia.
* Individuals with severe injuries or burns or limb amputation after breast surgery.
* Open wounds or infectious dermatitis on the oral and facial regions.
* Acute or infectious respiratory tract infections.
* Currently taking any medications.
* Respiratory therapy students.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Urinary salbutamol concentration | Urine samples will be collected at 30 minutes before nebulization, at 30 minutes, and 24 hours after nebulization.
  Quantitative measurement of salbutamol levels in urine samples at protocol-specified timepoints before and after nebulized bronchodilator administration using high performance liquid chromatography (HPLC).

SECONDARY OUTCOMES:
Heart rate | Heart rate will be recorded continuously from 5 minutes before, during, and 30 minutes, and after nebulization.
  Heart rate measured via continuous telemetry
Blood pressure | Blood pressure will be recorded from 5 minutes before, during, and 30 minutes after nebulization.
  Systolic and diastolic blood pressure
Saturation | Oxygen saturation will be recorded from 5 minutes before, during, and 30 minutes after nebulization.
  Oxygen saturation using a pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lin, PhD, Study Director — Chang Gung University; Li-Chun Chiu, MD, PhD, Principal Investigator — Linko Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lipworth BJ. Pharmacokinetics of inhaled drugs. Br J Clin Pharmacol. 1996 Dec;42(6):697-705. doi: 10.1046/j.1365-2125.1996.00493.x. PMID 8971424
- [Background] Dolovich MB, Dhand R. Aerosol drug delivery: developments in device design and clinical use. Lancet. 2011 Mar 19;377(9770):1032-45. doi: 10.1016/S0140-6736(10)60926-9. Epub 2010 Oct 29. PMID 21036392
- [Background] Yeo LY, Friend JR, McIntosh MP, Meeusen EN, Morton DA. Ultrasonic nebulization platforms for pulmonary drug delivery. Expert Opin Drug Deliv. 2010 Jun;7(6):663-79. doi: 10.1517/17425247.2010.485608. PMID 20459360
- [Background] Dhand R. New frontiers in aerosol delivery during mechanical ventilation. Respir Care. 2004 Jun;49(6):666-77. PMID 15165301
- [Background] Kern DG, Frumkin H. Asthma in respiratory therapists. Ann Intern Med. 1989 May 15;110(10):767-73. doi: 10.7326/0003-4819-110-10-767. PMID 2712460
- [Background] Christiani DC, Kern DG. Asthma risk and occupation as a respiratory therapist. Am Rev Respir Dis. 1993 Sep;148(3):671-4. doi: 10.1164/ajrccm/148.3.671. PMID 8368639
- [Background] Dimich-Ward H, Wymer ML, Chan-Yeung M. Respiratory health survey of respiratory therapists. Chest. 2004 Oct;126(4):1048-53. doi: 10.1378/chest.126.4.1048. PMID 15486362
- [Background] Dhand R. Intelligent nebulizers in the age of the Internet: The I-neb Adaptive Aerosol Delivery (AAD) system. J Aerosol Med Pulm Drug Deliv. 2010 Apr;23 Suppl 1(Suppl 1):iii-v. doi: 10.1089/jamp.2010.0818. No abstract available. PMID 20373913
- [Background] Denyer J, Dyche T. The Adaptive Aerosol Delivery (AAD) technology: Past, present, and future. J Aerosol Med Pulm Drug Deliv. 2010 Apr;23 Suppl 1(Suppl 1):S1-10. doi: 10.1089/jamp.2009.0791. PMID 20373904
- [Background] Chamberlain D, Kodgule R, Ganelin D, Miglani V, Fletcher RR. Application of semi-supervised deep learning to lung sound analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:804-807. doi: 10.1109/EMBC.2016.7590823. PMID 28324938
- [Background] Islam MA, Bandyopadhyaya I, Bhattacharyya P, Saha G. Multichannel lung sound analysis for asthma detection. Comput Methods Programs Biomed. 2018 Jun;159:111-123. doi: 10.1016/j.cmpb.2018.03.002. Epub 2018 Mar 9. PMID 29650306
- [Background] Messner E, Fediuk M, Swatek P, Scheidl S, Smolle-Juttner FM, Olschewski H, Pernkopf F. Multi-channel lung sound classification with convolutional recurrent neural networks. Comput Biol Med. 2020 Jul;122:103831. doi: 10.1016/j.compbiomed.2020.103831. Epub 2020 May 23. PMID 32658732
- [Background] Seren E. Frequency spectra of normal expiratory nasal sound. Am J Rhinol. 2005 May-Jun;19(3):257-61. PMID 16011131
- [Background] Sen I, Saraclar M, Kahya YP. A Comparison of SVM and GMM-Based Classifier Configurations for Diagnostic Classification of Pulmonary Sounds. IEEE Trans Biomed Eng. 2015 Jul;62(7):1768-76. doi: 10.1109/TBME.2015.2403616. Epub 2015 Feb 12. PMID 25700439
- [Background] Charleston-Villalobos S, Martinez-Hernandez G, Gonzalez-Camarena R, Chi-Lem G, Carrillo JG, Aljama-Corrales T. Assessment of multichannel lung sounds parameterization for two-class classification in interstitial lung disease patients. Comput Biol Med. 2011 Jul;41(7):473-82. doi: 10.1016/j.compbiomed.2011.04.009. Epub 2011 May 14. PMID 21571265
- [Background] Loeb M, McGeer A, Henry B, Ofner M, Rose D, Hlywka T, Levie J, McQueen J, Smith S, Moss L, Smith A, Green K, Walter SD. SARS among critical care nurses, Toronto. Emerg Infect Dis. 2004 Feb;10(2):251-5. doi: 10.3201/eid1002.030838. PMID 15030692
- [Background] Heinzerling A, Stuckey MJ, Scheuer T, Xu K, Perkins KM, Resseger H, Magill S, Verani JR, Jain S, Acosta M, Epson E. Transmission of COVID-19 to Health Care Personnel During Exposures to a Hospitalized Patient - Solano County, California, February 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):472-476. doi: 10.15585/mmwr.mm6915e5. PMID 32298249
- [Result] Denyer J, Prince I, Dixon E, Agent P, Pryor J, Hodson M. Evaluation of the Target Inhalation Mode (TIM) breathing maneuver in simulated nebulizer therapy in patients with cystic fibrosis. J Aerosol Med Pulm Drug Deliv. 2010 Apr;23 Suppl 1(Suppl 1):S29-36. doi: 10.1089/jamp.2009.0768. PMID 20373907
- [Result] Geller DE, Kesser KC. The I-neb Adaptive Aerosol Delivery System enhances delivery of alpha1-antitrypsin with controlled inhalation. J Aerosol Med Pulm Drug Deliv. 2010 Apr;23 Suppl 1(Suppl 1):S55-9. doi: 10.1089/jamp.2009.0793. PMID 20373910
- [Result] Nikander K, Prince I, Coughlin S, Warren S, Taylor G. Mode of breathing-tidal or slow and deep-through the I-neb Adaptive Aerosol Delivery (AAD) system affects lung deposition of (99m)Tc-DTPA. J Aerosol Med Pulm Drug Deliv. 2010 Apr;23 Suppl 1(Suppl 1):S37-43. doi: 10.1089/jamp.2009.0786. PMID 20373908
- [Result] Acharya J, Basu A. Deep Neural Network for Respiratory Sound Classification in Wearable Devices Enabled by Patient Specific Model Tuning. IEEE Trans Biomed Circuits Syst. 2020 Jun;14(3):535-544. doi: 10.1109/TBCAS.2020.2981172. Epub 2020 Mar 18. PMID 32191898